CLINICAL TRIAL: NCT07044999
Title: Evaluation of Balance and Physical Performance Under Dual Task Conditions in Individuals With and Without Generalized Joint Hypermobility
Status: Not yet recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH22
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hypermobility Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with hypermobility
  Interventions: Other: no intervention
- Control group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aims to evaluate balance and physical performance under dual task conditions in individuals with and without Generalized Joint Hypermobility (GJH), as determined by the Beighton score. All participants will undergo the One-Leg Stance Test and 30-Second Sit-to-Stand Test under both single-task (balance only) and dual-task (simultaneous cognitive task) conditions. The cognitive task will involve counting backward by sevens from a given number. Participants will also complete the Timed Up and Go (TUG) test under both single- and dual-task conditions. Additionally, the Berg Balance Scale (BBS) will be used for comprehensive balance assessment. Balance confidence will be evaluated using the Activities-specific Balance Confidence Scale (ABC-16), and fear of falling will be assessed with the Falls Efficacy Scale-International (FES-I). Changes in performance under dual-task conditions will be expressed as a percentage using the Dual Task Cost (DTC) formula

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years
* A Beighton score of 4 or higher (indicative of Generalized Joint Hypermobility)
* Willingness to participate in the study

Exclusion Criteria:

* Younger than 18 or older than 40 years
* Presence of neurological disorders (e.g., stroke, multiple sclerosis, peripheral neuropathy)
* History of vestibular system disorders (e.g., benign paroxysmal positional vertigo, vestibular neuritis)
* History of orthopedic conditions affecting the lower extremities (e.g., fracture, joint replacement, ligament injury)
* Cognitive impairment preventing the execution of cognitive tasks
* Diagnosis of systemic musculoskeletal diseases (e.g., rheumatoid arthritis, Ehlers-Danlos syndrome)
* Pregnancy
* Participation in balance training or neurological/physiotherapy programs within the last 6 months

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: hypermobile patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Performance in the One-Leg Stance Test | 0 day
  Assesses static balance capacity and the impact of a simultaneous cognitive task on postural control.
Performance in the 30-Second Sit-to-Stand Test | 0 day
  Evaluates lower extremity muscle endurance and functional strength under cognitive load
Performance in the Timed Up and Go (TUG) test | 0 day
  Measures dynamic balance, mobility, and the ability to maintain performance during divided attention.
Dual Task Cost (DTC) percentage | 0 day
  Quantifies the percentage change in performance when a cognitive task is added, reflecting dual-task interference.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS): | 0 day
  Provides a comprehensive evaluation of functional balance through various static and dynamic tasks. The maximum score is 56. Higher scores indicate that good balance.
Activities-specific Balance Confidence Scale (ABC-16) | 0 day
  Reflects the individual's perceived confidence in performing daily activities without losing balance.The maximum score is 100, the minimum score is 0. Higher scores indicate that high confidence patient's balance.
Falls Efficacy Scale-International (FES-I): | 0 day
  Assesses fear of falling during daily life activities, indicating fall-related psychological concerns. Higher scores indicate that high degree fear of falling